CLINICAL TRIAL: NCT03639779
Title: A Comparative Study of the Efficacy of Intralesional Sodium Thiosulfate Versus Intralesional Normal Saline for the Treatment of Dystrophic and Idiopathic Calcinosis Cutis, A Double-Blind Randomized Placebo-Controlled Trial
Brief Title: Efficacy of Intralesional Sodium Thiosulfate Versus Intralesional Saline for Dystrophic and Idiopathic Calcinosis Cutis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Time and resource constraints
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, David Weinstein, Assistant Professor of Dermatology, University of Central Florida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIO-18-14095
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Results first posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Calcinosis Cutis
Keywords: Calcinosis cutis; sodium thiosulfate; sodium chloride
MeSH Terms: conditions — Calcinosis Cutis | interventions — sodium thiosulfate; Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a parallel two-arm study comparing sodium thiosulfate and saline control.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sodium thiosulfate (Experimental): 50 ml vials of sodium thiosulfate (250mg/ml) will be used for treatment.
  Interventions: Drug: Sodium Thiosulfate
- Saline solution (Placebo Comparator): 30 ml vials of sodium chloride 0.9% will be used for the control treatment.
  Interventions: Other: Saline Solution

INTERVENTIONS:
Drug: Sodium Thiosulfate — A volume of 0.1 ml/cm2 of STS will be injected into each lesion.
  Arms: Sodium thiosulfate
Other: Saline Solution — A volume of 0.1 ml/cm2 of normal saline will be injected into the control lesion.
  Arms: Saline solution

SUMMARY:
The purpose of our research is to compare the effectiveness of 125mg/50ml sodium thiosulfate (STS) solution to normal saline (0.9% sodium chloride) when injected intralesionally for the treatment of calcinosis cutis. Our specific aim is to assess the response of dystrophic and idiopathic calcinosis cutis to the injections of sodium thiosulfate in our patients.

DETAILED DESCRIPTION:
Our specific aim is to assess the response of dystrophic and idiopathic calcinosis cutis to the injections of sodium thiosulfate in our patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult 18 years of age or older
* Must have health insurance will be eligible to participate
* Must have a current diagnosis of dystrophic or idiopathic calcinosis cutis
* Subjects must have at least 2 lesions of at least 2mm in size

Exclusion Criteria:

* Unable to read and speak English
* Allergy to any component of the sodium thiosulfate solution
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Women who are breastfeeding
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCF Health Lake Nona Office, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study had to be close early due to lack of support and time resulting in a lower number of participants than hoped for. 5 participants began the study, 1 was lost to follow-up. Each participant had 2 study lesions, each assigned to a different study arm.
Units Other Than Participants: Lesions
Groups:
- All Paticipants: All study participants received an injection of Sodium Thiosulfate into one lesion. They received an injection of saline in the control lesion
  50 ml vials of sodium thiosulfate (250mg/ml) were used for treatment. 30 ml vials of sodium chloride 0.9% will be used for the control treatment. A volume of 0.1 ml/cm2 of STS or normal will be injected into each lesion.
Period: Overall Study
Arm/Group | All Paticipants
Started | 5; 10 Lesions
Baseline | 5; 10 Lesions
Month 1 | 5; 10 Lesions
Month 2 | 4; 8 Lesions
Month 3 | 4; 8 Lesions
Completed | 4; 8 Lesions
Not Completed | 1; 2 Lesions
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All study participants received an injection of Sodium Thiosulfate into one lesion. They received an injection of saline in the control lesion.
Arm/Group | All Participants
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Lesion Size
Description: The lesion size is measured in square centimeters.
Time Frame: 3 months
Population: One participant was lost to follow up
Measure: Mean (Full Range); unit: cm^2
Arm/Group | Sodium Thiosulfate | Saline Solution
Number analyzed (Participants) | 5 | 5
cm^2
  Baseline | 2.8 [0.1 to 4] | 1.8 [0.4 to 4]
  3 Months: number analyzed (Participants) | 4 | 4
  3 Months | 3 [0 to 4] | 3.0 [0.1 to 4]

2. Primary Outcome: Physician Global Assessment (PGA)
Description: The PGA will be done by the physician to assess appearance and changes in the lesion. The lesion will be assigned a score from 0 (clear) to 4 (severe).
Time Frame: 3 months
Population: One participant was lost to follow up.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Sodium Thiosulfate | Saline Solution
Number analyzed (Participants) | 5 | 5
score on a scale
  Baseline | 4 [4 to 4] | 4 [4 to 4]
  3 Month: number analyzed (Participants) | 4 | 4
  3 Month | 3 [0 to 4] | 3.25 [1 to 4]

3. Primary Outcome: Visual Analog Scale (VAS) for Pain
Description: The VAS for pain is used to assess the pain associated with the lesion. The pain will be recorded as a number from 1 (no pain) to 10 (severe pain).
Time Frame: 3 months
Population: One participant was lost to follow up.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Sodium Thiosulfate | Saline Solution
Number analyzed (Participants) | 5 | 5
score on a scale | 3.6 [0.4 to 10] | 2.6 [0 to 6.6]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Sodium Thiosulfate | Saline Solution
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

LIMITATIONS AND CAVEATS:
The study had to be closed early due to lack up support/resources.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-15): https://cdn.clinicaltrials.gov/large-docs/79/NCT03639779/Prot_SAP_002.pdf
  • Informed Consent Form (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT03639779/ICF_003.pdf